CLINICAL TRIAL: NCT02440178
Title: Phase II Trial of Micafungin Prophylaxis During Induction Chemotherapy for Patients With Acute Leukemia
Brief Title: Micafungin Prophylaxis During 1st Induction Chemotherapy for De Novo Acute Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNUH-micafungin
Record Dates: First submitted 2015-05-03; First posted 2015-05-12 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2017-10

CONDITIONS: Acute Leukemia
Keywords: leukemia; induction; prophylaxis; antifungal; micafungin; phase II
MeSH Terms: conditions — Leukemia | interventions — Micafungin

ARMS (1):
- micafungin prophylaxis (Experimental): Patients received 50 mg micafungin intravenously once daily from the initiation of induction chemotherapy to recovery of neutrophil count (absolute neutrophil count > 500/μg for three consecutive days), suspected fungal infection, or occurrence of drug-related toxicity.
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin
  Other Names: mycamine

SUMMARY:
The purpose of this study is to determine whether prophylaxis with micafungin is effective in the induction chemotherapy for newly diagnosed acute leukemia patients.

DETAILED DESCRIPTION:
Medically fit patients with newly diagnosed acute leukemia received 50 mg micafungin intravenously once daily from the initiation of first induction chemotherapy to recovery of neutrophil count, suspected fungal infection, or unacceptable drug-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

A. patients belong to either A-1 or A-2 A-1. patients with newly diagnosed acute myeloid leukemia who approve to get induction chemotherapy with (cytarabine plus idarubicin) or (modified Fludarabine + cytarabine + idarubicin ) A-2. patients with newly diagnosed acute lymphoid leukemia who approve to get induction chemotherapy with VPDL (vincristine + prednisolone + daunorubicin + L-asparaginase), C-VPDL (cyclophosphamide + vincristine + prednisolone + daunorubicin + L-asparaginase), or (R)-hyperCVAD ((Rituximab) + cyclophosphamide + vincristine + Adriamycin + dexamethasone) B. Eastern Cooperative Oncology Group performance status score is equal to or more than 2 C. patients who voluntarily sign the agreement

Exclusion Criteria:

A. evidence of proven/probable/possible fungal infection within 30 days before induction chemotherapy B. hypersensitivity to echinocandin C. patients had other malignancy within 5 years D. previous treatment history with chemotherapy, radiation therapy, or immunosuppressive therapy.

E. pregnant or breast-feeding women F. immunodeficient patients including AIDS G. patients with uncontrolled seizure or psychiatric disorder H. clinically significant heart disorder (myocardial infarction within 3 months or left ventricular ejection fraction < 40%) I. interstitial lung disease J. previous organ transplantation history K. galactose intolerance L. patients who participated this study before.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-09-19 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, Dr., Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Park H, Youk J, Shin DY, Hong J, Kim I, Kim NJ, Lee JO, Bang SM, Yoon SS, Park WB, Koh Y. Micafungin prophylaxis for acute leukemia patients undergoing induction chemotherapy. BMC Cancer. 2019 Apr 16;19(1):358. doi: 10.1186/s12885-019-5557-9. PMID 30991992

RESULTS

PARTICIPANT FLOW:
Groups:
- Micafungin Prophylaxis: 50 mg micafungin intravenously once daily from the initiation of induction chemotherapy to recovery of neutrophil count (absolute neutrophil count > 500/μg for three consecutive days), suspected fungal infection, or occurrence of drug-related toxicity
Period: Overall Study
Arm/Group | Micafungin Prophylaxis
Started | 66
Completed | 46
Not Completed | 20

BASELINE CHARACTERISTICS:
Groups:
- Micafungin Prophylaxis: The baseline characteristics of total patients
Arm/Group | Micafungin Prophylaxis
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 57
  >=65 years | 7
Age, Continuous [Median (Full Range); unit: years] | 51 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 65
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Proven/Probable/Possible Invasive Fungal Infection
Description: proven fungal infection: proven by positive culture for fungus with symptoms and signs of a fungal infection probable fungal infection: direct or indirect detection (galactomannan antigen or serum β-D-glucan) with clinical and radiographic findings possible fungal infection: sufficient clinical evidence for fungal infection was present without mycological evidence
Time Frame: the day of 6 weeks after induction chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Micafungin Prophylaxis: The outcomes of fungal infections
Arm/Group | Micafungin Prophylaxis
Number analyzed (Participants) | 65
Participants
  Proven fungal infection | 1
  Probable fungal infection | 0
  Possible fungal infection | 2
  Non fungal infection | 62

2. Secondary Outcome: Overall Survival
Description: The survival of patients till 12 weeks after induction chemotherapy
Time Frame: the day of 12 weeks after induction chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Survival Outcome: The survival of patients till 12 weeks after induction chemotherapy
Arm/Group | Survival Outcome
Number analyzed (Participants) | 65
Participants
  survival | 62
  death | 3

3. Secondary Outcome: Non-relapse Mortality
Description: The outcomes of non-relapse mortality: The incidence of death without a previous relapse or progression
Time Frame: The day of 12 weeks after induction chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Non-relapse Mortality: Non-relapse mortality was defined as the incidence of death without a previous relapse or progression.
Arm/Group | Non-relapse Mortality
Number analyzed (Participants) | 65
Participants
  Non-relapse mortality | 3
  survival | 62

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Adverse Events: Serious adverse events: life-threatening adverse events Other adverse events: non-serious adverse events during treatment
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 3/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 3/65
OTHER ADVERSE EVENTS (reported when occurring in more than 4.6% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events (N=65)
Liver function test abnormality (Hepatobiliary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02440178/Prot_SAP_ICF_000.pdf